CLINICAL TRIAL: NCT04007926
Title: Effects of Exercise Training on Insulin Sensitivity in South Asians at Risk of Diabetes: the Roles of Skeletal Muscle Microvasculature and Mitochondrial Metabolism
Brief Title: Mechanisms of Insulin Resistance and Exercise in South Asians
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: University of Glasgow (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Professor Jason Gill, Professor, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 265320
Record Dates: First submitted 2019-06-28; First posted 2019-07-05 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Insulin Resistance
Keywords: insulin resistance; aerobic exercise; resistance exercise; exercise training; South Asians
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Masking Description: Masking is not possible due to nature of intervention (exercise training programme).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Participants assigned to the control arm of the study will be asked to maintain their normal dietary and exercise habits.
- Aerobic exercise group (Experimental): Participants randomised to the aerobic exercise intervention will undertake a 12-week aerobic exercise training programme.
  Interventions: Behavioral: Aerobic exercise programme
- Resistance exercise group (Experimental): Participants randomised to the resistance exercise intervention will undertake a 12-week aerobic exercise training programme.
  Interventions: Behavioral: Resistance exercise programme

INTERVENTIONS:
Behavioral: Aerobic exercise programme — Participants will start with 3 x 20 minute exercise sessions in the first week, building up to 5 x 60 minutes of exercise by weeks 9-12 of the intervention, at an intensity of 65-80% of predicted maximum heart rate.
  Arms: Aerobic exercise group
Behavioral: Resistance exercise programme — Participants will undertake two supervised sessions per week. The exercises performed during each session will consist of leg press, calf press, leg extension, leg curl, chest press, shoulder press, lateral pull down and seated row. Exercises will be performed at 60-80% 1RM. In weeks 1-2 participants will perform, during each session, a single set of 5-10 repetitions of each exercise (tiring but comfortably achievable) to ensure they are comfortable with the exercises and are performing these in the correct form. In weeks 3-4 participants will perform, during each session, two sets of each exercise to voluntary muscular failure - defined as not being able to perform single another repetition. In weeks 5-12 this will progress to 3 sets of each exercise to voluntary muscular failure, in each session.
  Arms: Resistance exercise group

SUMMARY:
This study determines the effect of aerobic and resistance exercise training on whole-body and skeletal muscle insulin sensitivity in south Asians and evaluate the mechanisms which contribute to improvements in insulin sensitivity after exercise training.

DETAILED DESCRIPTION:
South Asians (SA) have 2-4 fold higher risk of type 2 diabetes and develop the disease at lower body weights and younger ages than white Europeans. Lower cardiorespiratory fitness and capacity for muscle fat oxidation contributes substantially to SAs' greater insulin resistance, the extent to which this can be improved by exercise training is unclear. This randomised controlled trial will investigate the effects of a 12-week aerobic or resistance exercise training intervention on insulin sensitivity (hyperinsulinaemic-euglycaemic clamp) in South Asian adults (22 control, 22 aerobic exercise group and 22 resistance exercise group). The study will also explore the mechanisms within skeletal muscle which mediate these changes by evaluating aerobic and resistance exercise-training induced changes: in basal and insulin-stimulated microvascular blood volume (using contrast-enhanced ultrasound); skeletal muscle mitochondrial function; and lipid droplet morphology and spatial interaction with mitochrondria, muscle fibre capillarisation, endothelial content of key enzymes controlling dilation/constriction and GLUT-4 translocation (using confocal immunofluorescence microscopy and transmission electron microscopy methods). Thus, this work will integrate physiological and molecular data to determine the extent to which exercise training can improve insulin sensitivity in SA and the mechanisms underpinning this improvement. This knowledge is important for optimising diabetes prevention interventions in SAs and identification of potential novel therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Male
* South Asian ethnicity (self-report of both parents of Indian, Pakistani, Bangladeshi or Sri Lankan origin)
* Age 30-65 years
* At least 10% 10-year risk of developing type 2 diabetes, determined using the QDiabetes®2018 risk score (http://qdiabetes.org/2018/index.php)

Exclusion Criteria:

* Female
* Diabetes (physician diagnosed or HbA1c ≥48 mmol/mol on screening)
* History of cardiovascular disease
* Hypertension (taking anti-hypertensives or BP consistently ≥ 150/90 mmHg on screening).
* Regular participation in vigorous physical activity
* Regular participation in resistance exercise
* Current smoking
* Taking drugs or supplements thought to affect carbohydrate or lipid metabolism
* Taking drugs affecting blood clotting (e.g. aspirin)
* Current treatment with anti-obesity drugs
* Any other significant illness that would prevent full participation in the study

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Whole-body Insulin sensitivity | Change between baseline and 12 weeks.
  Change in whole-body insulin sensitivity measured by hyperinsulinaemic-euglycaemic clamp.

SECONDARY OUTCOMES:
Insulin-stimulated GLUT4 translocation | Change between baseline and 12 weeks.
  Change in insulin-stimulated GLUT4 translocation in muscle biopsies from vastus lateralis using immunofluorescence microscopy
Microvascular blood volume | Change between baseline and 12 weeks.
  Change in fold-increase in insulin stimulated quadriceps muscle blood volume measured using contrast enhanced ultrasound.
Muscle mitochondrial function | Change between baseline and 12 weeks.
  Change in mitochondrial function (oxygen consumption rate) in isolated skeletal muscle mitochondria from the vastus lateralis measured using respirometry
Lipid droplet content in skeletal muscle | Change between baseline and 12 weeks.
  Change in fibre type-specific (type 1 and type 2) and subcellular-specific (subsarcolemmal and intermyofibrillar) lipid droplet content in muscle biopsies from vastus lateralis using immunofluorescence microscopy
Lipid droplet proximity to mitochondria in skeletal muscle | Change between baseline and 12 weeks.
  Change in proportion of lipid droplets in contact with mitochondria in subsarcolemmal and intermyofibrillar compartments of type 1 and type 2 muscle fibres in muscle biopsies from vastus lateralis using immunofluorescence microscopy
Microvascular density in skeletal muscle | Change between baseline and 12 weeks.
  Change in fibre-type specific capillarisation in muscle biopsies from vastus lateralis
Change in enzymes controlling insulin-mediated increases in perfusion in skeletal muscle | Change between baseline and 12 weeks.
  Change in endothelial specific protein content and phosphorylation of key microvascular enzymes in muscle biopsies from vastus lateralis assessed using quantitative immunofluorescence.
Maximal oxygen uptake | Change between baseline and 12 weeks.
  Change in maximal oxygen uptake consumption assessed using continuous incremental uphill walking protocol until volitional exhaustion.
Muscle maximal voluntary contraction | Change between baseline and 12 weeks.
  Change in knee extensor muscles maximal voluntary contraction
Lower body muscle strength | Change between baseline and 12 weeks.
  Change in 1-RM (one maximal repetition) (kg) for leg press.
Upper body muscle strength | Change between baseline and 12 weeks.
  Change in 1-RM (one maximal repetition) (kg) for chest press.
Grip strength | Change between baseline and 12 weeks.
  Change in grip strength (kg).
Fat mass | Change between baseline and 12 weeks.
  Change in fat mass measured with bioelectrical impedance analysis (BIA).
Fat-free mass | Change between baseline and 12 weeks.
  Change in fat-free mass measured with bioelectrical impedance analysis (BIA).
Weight | Change between baseline and 12 weeks.
  Change in weight (kg).
Waist circumference | Change between baseline and 12 weeks.
  Change in waist circumference (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Gill, PhD, Principal Investigator — University of Glasgow
Locations (1):
- University of Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marx N, Davies MJ, Grant PJ, Mathieu C, Petrie JR, Cosentino F, Buse JB. Guideline recommendations and the positioning of newer drugs in type 2 diabetes care. Lancet Diabetes Endocrinol. 2021 Jan;9(1):46-52. doi: 10.1016/S2213-8587(20)30343-0. Epub 2020 Nov 4. PMID 33159841